CLINICAL TRIAL: NCT06399835
Title: Comparing Enavogliflozin and Pioglitazone as Add-ons to Metformin With/Without Dipeptidyl Peptidase-4 Inhibitors in Type 2 Diabetes
Brief Title: Enavogliflozin vs. Pioglitazone on Glucose and Atherosclerosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2310-859-002
Record Dates: First submitted 2024-04-26; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin (Experimental): Enavogliflozin 0.3 mg
  Interventions: Drug: Enavogliflozin
- Pioglitazone (Active Comparator): Pioglitazone 15 mg
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Enavogliflozin — Enavogliflozin 0.3mg once daily
  Other Names: Envlo Tab.
  Arms: Enavogliflozin
Drug: Pioglitazone — Pioglitazone 15mg once daily
  Other Names: Actos Tab.
  Arms: Pioglitazone

SUMMARY:
The current study aimed to thoroughly compare a thiazolidinedione and an sodium-glucose cotransporter-2 (SGLT2) inhibitor regarding various clinical issues including atherosclerosis. Enavogliflozin is compared to Pioglitazone in the glucose-lowering effects of adding to the treatment of patients with type 2 diabetes whose HbA1c levels are not controlled by Metformin with or without DPP-4 inhibitors. Additionally, the study will compare changes in other metabolic or cardiovascular risk factors, such as triglycerides, high density lipoprotein cholesterol (HDLc), uric acid, blood pressure, and inflammatory markers, between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with a glycated hemoglobin (HbA1c) level of 7.0 - 10.5% at screening
* Males or females aged 20-80 years
* Individuals who have been taking Metformin (≥ 500mg) with or without a DPP-4 inhibitor (such as Sitagliptin, Vildagliptin, Saxagliptin, Linagliptin, Gemigliptin, Alogliptin, Teneligliptin, Anagliptin, Evogliptin) for at least the past 3 months
* Body mass index ≥ 23 kg/m²
* Estimated glomerular filtration ratio (eGFR) ≥ 60 ml/min/1.73m²

Exclusion Criteria:

* Patients with Type 1 Diabetes, Gestational Diabetes, or secondary diabetes due to other causes
* Patients with a history of acute cardiovascular disease within the last 3 months prior to the screening visit
* Pregnant or breastfeeding patients, or patients not using contraception. Patients with chronic Hepatitis B or C (excluding healthy carriers of Hepatitis B), or liver disease (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal)
* Patients with heart failure or a history of heart failure
* Individuals with a history of cancer within the past 5 years (excluding those adequately treated for squamous cell carcinoma or thyroid cancer)
* Patients who have participated in another clinical study within the last 30 days
* Alcohol addiction
* Patients for whom the use of Enavogliflozin or Pioglitazone is contraindicated
* Patients taking other oral hypoglycemic agents or insulin or other investigational drugs
* Patients deemed unsuitable for the study based on the investigator's judgment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of HbA1c from the baseline | 24 weeks

SECONDARY OUTCOMES:
Patients achieving HbA1c levels below 7% | 24 weeks
  N and percentage of the patients
Changes of body fat (whole body fat, abdominal fat) | 24 weeks
  kg, %; measured with bioelectrical impedance analysis
Changes of body weight | 12 weeks, 24 weeks
Changes of glucose levels (fasting, 2-hour postprandial) | 12 weeks, 24 weeks
  mg/dL
Changes of systolic/diastolic blood pressures | 12 weeks, 24 weeks
  mmHg
Changes of lipids (total cholesterol, HDLc, low density lipoprotein cholesterol [LDLc], triglycerides) | 12 weeks, 24 weeks
  mg/dL
Changes of electrolytes (uric acid) | 12 weeks, 24 weeks
  mg/dL
Changes in parathyroid hormone | 12 weeks, 24 weeks
  pg/mL
Changes in 25-hydroxyl vitamin D3 | 12 weeks, 24 weeks
  ng/mL
Changes of albuminuria | 12 weeks, 24 weeks
  mg/g
Changes of urine electrolytes (Na, K, Cl, Ca, P, glucose) | 12 weeks, 24 weeks
  mg/dL
Changes in ketone body | 12 weeks, 24 weeks
  umol/L
Changes of carotid intima-media thickness | 24 weeks
  maximal thickness (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, M.D. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No